CLINICAL TRIAL: NCT03626129
Title: Randomised Comparison of Oximetry Guided Deflation Versus Traditional Rapid Deflation When Removing the TR-band After Radial Angiography or Angioplasty The Access-III Study
Brief Title: Oximetry Guided Versus Traditional Rapid Deflation Technique for Achieving Hemostasis After Radial Procedures
Acronym: ACCESS-III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Terumo Corporation (Industry)
Responsible Party: Principal Investigator, Christian Juhl Terkelsen, MD, DmSc, PhD, Associate professor, Aarhus University Hospital Skejby
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-159-18
Record Dates: First submitted 2018-08-01; First posted 2018-08-10 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Radial Artery
Keywords: Haemostasis; Trans radial band; Coronary angiography; Radial artery occlusion; Percutaneous coronary intervention
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional rapid deflation (No Intervention): Group A: At time of sheath removal 15 ml. air is inflated in the TR-band. The sheath is removed. Air is deflated until bleeding, and 1-2 ml. air is then re-inflated to achieve hemostasis, and the volume air inflated is registered ("Initial inflated air volume"). Every 20 minutes 1/3 of the initial inflated air volume is deflated. If bleeding occurs then air is re-inflated until hemostasis and then additional 1-2 ml. air is inflated. This routine is repeated until hemostasis is achieved (TR-band fully deflated without bleeding).
- Oximetry guided deflation (Experimental): Group B: Initial step with sheath removal as in group A. Before departure from the cath.lab. a "Patent hemostasis test" (see description in "Interventions" below) is performed. Further action as described in "Interventions" below.
  Interventions: Procedure: Oximetry guided deflation

INTERVENTIONS:
Procedure: Oximetry guided deflation — At the cath.lab. (Step 1) a hemostasis test is performed: oxymetry device on the thumb, compress a.ulnaris, evaluate if curve on device (="Patent hemostasis"). If patent no further action. If not patent, air is deflated until a.radialis is patent (curve on device and no bleeding). If bleeding occurs before patency then re-inflate 1-2 ml. air until hemostasis (="no patent hemostasis"). In patients with "Patent hemostasis" no action is taken in sixty minutes whereafter the TR-band is fully deflated (Step 2), and if bleeding then air is re-inflated until hemostasis and step 2 is repeated every 20 minutes until the TR-band is fully deflated with hemostasis. If "no patent hemostasis" at cath.lab. a hemostasis test is performed after 20 min. If "patent hemostasis" is achieved no action is taken in sixy minutes (as above). If still "not patent" then further action as in group A.
  Arms: Oximetry guided deflation

SUMMARY:
After performing a radial angiography/percutaneous coronary intervention (CAG/PCI), the sheath is removed and a compression device is used to achieve hemostasis. Recent studies have indicated that rapid deflation techniques resulting in early removal of the compression device is associated with a low incidence of radial artery occlusion (RAO).

The purpose of the present study is to evaluate whether an even faster removal of the compression device can be achieved if using oximetry guided rapid deflation compared to traditional rapid deflation, and whether this is associated with a lower incidence of RAO.

DETAILED DESCRIPTION:
3600 patients are randomized 1:1 to a traditional rapid deflation technique (Group A) versus an oximetry guided rapid deflation technique (Group B).

Before randomisation between the two deflation techniques French size of the sheath is chosen. If the operator has a preference for the size of the sheath then this size is used (5F/6F, estimated N=1200). If the operator has no preference for the size of the sheath then patients are randomized between 5 and 6 French sheath (N=2400).

Randomization between traditional rapid deflation technique (Group A) versus oximetry guided rapid deflation technique (Group B) is then stratified according to French size of the sheath used (5 French, 6 French). Terumo Glidesheath Slender is routinely used in both arms.

Assuming that the incidence of RAO (Barbeau type D, see below) can be reduced from 1.5% to 0.5% a total of 1547 patients are needed in each group if using an alfa=0.05 and beta 0.80. Assuming that the incidence of RAO or subocclusion (Barbeau type C or D, see below) can be reduced from 4% to 2% a total of 1141 patients are needed in each group to document this difference if using an alfa=0.05 and beta 0.80. The investigators plan to randomize 1800 in each group comparing oximetry guided rapid deflation with traditional rapid deflation. Assuming that the time from sheath removal to transradial-band (TR-band) removal (hemostasis) is 125 minutes with the traditional rapid deflation technique, and 110 minutes with the oximetry guided deflation technique, and the standard deviation is 60 minutes, then a total number of 253 patients are needed in each group to document a possible difference.

Data are analyzed by the intention-to-treat principle.

4-5 centres are expected to include patients.

Oral and written informed consent is collected at the ward or in the Cath.lab. The informed consent is signed before intervention.

Included patient can withdraw their assignment from the study at any time without consequence

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for radial angiography or angioplasty.
* Patients with normal flow in a.ulnaris before the procedure (Barbeau type A or B).
* Age > 18 years.
* Patients able to cooperate and understand information given by the hospital staff.

Exclusion Criteria:

* Patients not able to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3600 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
RAO (Reverse Barbeau type D) during index hospitalisation | Day 1 (Evaluated at time of TR-band removal)
  The reverse Barbeau involves compression of the ulnar artery and evaluation of the radial oximetric waveform. This documents the flow through the radial artery post-hemostasis, were a test result A is an open artery and D is an occluded artery.
Time from sheath removal to removal of the TR-band | Day 1
  The time period will be recorded in the cath. lab. and in the ward.
Proportion who have the TR-band removed within 90,120 and 180 minutes | Day 1
  Calculated with STATA, statistical software
RAO (Reverse Barbeau type D) at follow-up | After 1 month
  The reverse Barbeau involves compression of the ulnar artery and evaluation of the radial oximetric waveform. This documents the flow through the radial artery post-hemostasis, were a test result A is an open artery and D is an occluded artery.

SECONDARY OUTCOMES:
RAO or subocclusion during index hospitalisation | Day 1 (Evaluated at time of TR-band removal)
  Evaluated by reverse Barbeau Test (type C+D) were a test result A is an open artery and D is a occluded artery and hence B + C are a subocclusion.
Hematoma > 2.5 cm | Day 1 (Evaluated at time of discharge)
  Development of hematoma is monitored at the ward at time of discharge.
Time from sheath removal to discharge | Day 1
  The discharge time is recorded in the patient file
Discomfort in the arm | At 1 month and 3 months
  The pain numeric rating scale (NRS), on which patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain")
RAO or subocclusion at follow-up | At 1 month
  Evaluated by reverse Barbeau Test (type C+D) were a test result A is an open artery and D is a occluded artery and hence B + C are a subocclusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of cardiology, Aarhus University Hospital in Skejby, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No